CLINICAL TRIAL: NCT06797310
Title: Evaluating the Effectiveness and Tolerance of Baricitinib in the Treatment of Acute Alopecia Areata With Active Hair Shedding: A Prospective Open-Label Study
Acronym: MQ7422
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, National Taiwan University Clinical Trial Center, Sung-Jan Lin, National Taiwan University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202401193MIPB
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Alopecia Areata
Keywords: Acute alopecia areata; active hair shedding
MeSH Terms: conditions — Alopecia Areata | interventions — baricitinib

STUDY DESIGN:
Intervention Model Description: Prospective open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Baricitinib Treatment for Acute Alopecia Areata with Active Hair Shedding (Experimental): This study arm evaluates the effectiveness of baricitinib in patients with acute alopecia areata (AA) experiencing active hair shedding. Participants will receive baricitinib at a dose of 4 mg once daily for 16 weeks. Patients who achieve the primary endpoint, defined as an iSARS-AA score of 20 or less at week 16, will taper to 2 mg once daily for an additional 16 weeks before discontinuation. The intervention aims to rapidly halt hair shedding and promote regrowth, with follow-up visits scheduled at weeks 0, 4, 8, 12, 16, 24, 32, 36, 44, and 52 to monitor treatment response and potential relapse.
  Interventions: Drug: Baricitinib

INTERVENTIONS:
Drug: Baricitinib — This study evaluates the use of baricitinib 4 mg once daily for 16 weeks in patients with acute alopecia areata (AA) experiencing active hair shedding. Unlike prior studies focusing on chronic AA with extensive hair loss (SALT ≥ 50), this intervention targets the acute phase, aiming to halt shedding within 4-6 weeks-faster than conventional treatments like corticosteroids. Patients meeting the primary endpoint (iSARS-AA ≤ 20 at week 16) will taper to 2 mg daily for an additional 16 weeks. Scheduled follow-ups at weeks 0, 4, 8, 12, 16, 24, 32, 36, 44, and 52 ensure comprehensive monitoring, distinguishing this study from others with shorter follow-ups or less frequent assessments.

SUMMARY:
Alopecia areata (AA) in the acute phase with active hair shedding causes significant psychological distress, prompting the need for effective treatment. While baricitinib has shown efficacy in chronic AA with extensive hair loss (SALT ≥ 50), its impact on acute AA remains unclear. Clinical observations suggest that baricitinib can reduce or halt hair shedding within 4-6 weeks, offering a faster response than conventional treatments like systemic corticosteroids. This 16-week, single-center, open-label study aims to evaluate the effectiveness of baricitinib in 30 patients with acute AA and active shedding. Participants will receive 4 mg daily for 16 weeks, with responders tapering to 2 mg for an additional 16 weeks. Follow-up visits will occur at weeks 0, 4, 8, 12, 16, 24, 32, 36, 44, and 52. The primary endpoint is achieving an iSARS-AA score of 20 or less at week 16. This study will provide real-world insights into baricitinib's role in managing acute AA.

DETAILED DESCRIPTION:
Alopecia areata (AA) patients in the acute phase with active hair shedding experience significant psychological distress and an urgent need for effective treatment. The autoimmune nature of AA, driven by T-cell-mediated attacks on anagen hair follicles, leads to progressive hair loss. While baricitinib has been shown to promote hair regrowth in chronic AA with extensive hair loss (SALT ≥ 50), its efficacy in acute AA with active shedding has not been evaluated in BRAVE-AA1/2 trials. Clinical observations suggest that baricitinib can reduce or halt hair shedding within 4-6 weeks, offering a faster response compared to conventional treatments such as systemic corticosteroids, which often take longer or fail to achieve this outcome. This study aims to evaluate the effectiveness of baricitinib in patients with acute AA experiencing active shedding in a real-world setting. A 16-week, single-center, open-label, prospective trial will be conducted, enrolling 30 patients with active AA and progressive hair loss. Participants will receive 4 mg of baricitinib daily for 16 weeks, with responders tapering to 2 mg for an additional 16 weeks before discontinuation. Scheduled follow-up visits will be conducted at weeks 0, 4, 8, 12, 16, 24, 32, 36, 44, and 52. The primary endpoint is achieving an iSARS-AA score of 20 or less at week 16. Findings from this study will provide valuable insights into the real-world effectiveness of baricitinib in managing acute AA with active hair shedding.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be between 18 and 65 years of age (inclusive) at the time of enrollment. Subjects are eligible if they are male or nonpregnant, nonbreastfeeding female patients.
2. Active AA is defined as 30% or more of scalp surface area with active shedding via pull test
3. Current AA episode onset within 3 months

Exclusion Criteria:

1. Causes of acute hair shedding other than AA;
2. AA, in which the activity and/or onset time cannot be accurately determined;
3. Other medical concomitant conditions that require the use of systemic corticosteroids or immunosuppressants within 8 weeks of the baseline visit;
4. Intralesional steroid injection for AA within 4 weeks;
5. Previous treatment with oral JAKi with an inadequate response;
6. Have evidence of active TB or latent TB without completing at least 4 weeks of appropriate treatment;
7. Have any of the following specific abnormalities on screening laboratory tests: ANC <1,000 cells/mm³; ALC <500 cells/mm³; Hb levels <8 g/dL, platelets <100,000 cells/μL; AST or ALT ≥2 × ULN; ALP ≥2 × ULN; TBL ≥1.5 × ULN; eGFR <60 mL/min/1.73m2
8. Have an active, serious infection, including localized infection;
9. Have had symptomatic herpes zoster infection within 12 weeks before randomization. Have a history of disseminated/complicated herpes zoster (for example, ophthalmic zoster or CNS involvement);
10. Have a positive test for hepatitis B virus (HBV) infection, defined as positive for hepatitis B surface antigen (HBsAg), or positive for hepatitis B core antibody (HBcAb) and positive HBV deoxyribonucleic acid (DNA).
11. Have hepatitis C virus (HCV) infection (hepatitis C antibody-positive and HCV ribonucleic acid [RNA]-positive);
12. Have evidence of HIV infection and/or positive HIV antibodies;
13. Have been exposed to a live vaccine within 12 weeks or are expected to need/receive a live vaccine during the course of the study (except herpes zoster vaccination);
14. Have a history of chronic alcohol abuse, intravenous drug abuse, or other illicit drug abuse within the 2 years before study entry;
15. Have a history of cancer, or have an active primary or recurrent malignant disease; or have been in remission from clinically significant malignancy for <5 years (except fully treated NMSC and SCCis of the cervix). Have a history of lymphoproliferative disease; have signs or symptoms suggestive of possible lymphoproliferative disease, including lymphadenopathy or splenomegaly;
16. Have experienced any of the following within 12 weeks of screening: VTE (DVT/pulmonary embolism [PE]), myocardial infarction (MI), unstable ischemic heart disease, stroke, or New York Heart Association Stage III/IV heart failure;
17. Have had any major surgery within 8 weeks before screening or will require major surgery during the study that, in the opinion of the investigator would pose an unacceptable risk to the patient;
18. Have a history or presence of cardiovascular, respiratory, hepatic, gastrointestinal, endocrine, hematological, neurological, or neuropsychiatric disorders or any other serious and/or unstable illness that in the opinion of the investigator, could constitute an unacceptable risk when taking the investigational product or interfere with the interpretation of data;
19. Any other condition in the opinion of the investigator which would interfere with the study assessments or procedure.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-23 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure is the iSARS-AA (International Alopecia Areata Research Society - Alopecia Areata Severity Score) | From enrollment to the end of treatment at 8 weeks
  The primary outcome measure is the iSARS-AA (International Alopecia Areata Research Society - Alopecia Areata Severity Score), with the goal of achieving a score of 20 or less at week 16. This outcome will assess the reduction in alopecia severity and the effectiveness of baricitinib in halting active hair shedding in patients with acute alopecia areata.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No